CLINICAL TRIAL: NCT07097558
Title: The Effect of Mandala Coloring and Music Listening on Premenstrual Syndrome Symptoms and Quality of Life: A Randomized Controlled Trial
Brief Title: Mandala and Music for PMS Relief
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Rukiye Duman, RESEARCH ASSISTANT, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulUC-EBE-RD-01
Record Dates: First submitted 2025-07-25; First posted 2025-07-31 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Mandala Coloring; Music Listening; Premenstrual Syndrome-PMS
Keywords: Music Listening; music; art therapy; mandala coloring; Premenstrual Syndrome
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study includes a mandala coloring group, a music performance group, and a control group. Participating students will be informed about the study and provided with an "Informed Consent Form" and a "Voluntary Consent Form." The mandala painting intervention will be administered twice a week for 8 weeks to the mandala painting group, and the music performance will be administered twice a week for 30 minutes, twice a day, for 8 weeks. Participants in the music performance group will listen to classical music. The control group will not receive any intervention. Data will be collected using a "Personal Information Form," the "Premenstrual Syndrome Scale (PMSS)," and the "WHOQOL-BREF-TR Quality of Life Scale."
Who Masked: Participant
Masking Description: To determine the groups for university students who meet the sampling criteria for the study's randomization, participants will be assigned to the experimental and control groups using the "Randomizer.org" program. Numbers 1 to 120 will be randomized into three groups using a computer-assisted randomization program (https://www.randomizer.org). Students in the experimental and control groups will be prevented from interacting with each other to avoid being affected by the interventions. Inclusion and exclusion criteria, as well as exclusion from the study during the study, are specified below.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mandala coloring group (Experimental): The mandala painting intervention will be administered twice a week for 8 weeks for the mandala painting group.
  Interventions: Other: Mandala coloring group
- Music listening group (Experimental): The music listening group will listen to classical music twice a week for 8 weeks for 30 minutes, twice a day.
  Interventions: Other: Music listening group
- Control group (Experimental): The control group will not receive any intervention.
  Interventions: Other: control group

INTERVENTIONS:
Other: Mandala coloring group — The mandala painting intervention will be administered twice a week for 8 weeks for the mandala coloring group.
  Arms: Mandala coloring group
Other: Music listening group — The music listening group will listen to classical music twice a week for 8 weeks for 30 minutes, twice a day.
  Arms: Music listening group
Other: control group — The control group will not receive any intervention.
  Arms: Control group

SUMMARY:
Purpose: The aim of this project is to examine the effects of mandala painting and music performance interventions on premenstrual syndrome symptoms and quality of life.

The hypotheses of the study are as follows:

Coloring mandalas has a positive effect on premenstrual syndrome symptoms. Listening to music has a positive effect on premenstrual syndrome symptoms. Listening to music has a positive effect on quality of life. Coloring mandalas has a positive effect on quality of life.

DETAILED DESCRIPTION:
Purpose: The aim of this project is to examine the effects of mandala painting and music performance interventions on premenstrual syndrome symptoms and quality of life.

The study aims to reach all students experiencing PMS symptoms without resorting to sample calculations. Therefore, because a high effect size is expected in the study, a Cohen's standard effect size of 0.70, which is between medium and large, was assumed. Therefore (α = 0.05, effect size = 0.70, 1-β = 0.80), the minimum sample size was calculated as 120 participants (n = 40 for each group).

The study included a mandala painting group, a music performance group, and a control group. The mandala painting intervention will be administered twice a week for 8 weeks, and the music performance will be administered twice a week for 30 minutes, twice a day, for 8 weeks. Participants in the music performance group will listen to classical music. The control group will not receive any intervention. At the beginning of the study, data will be collected using a Personal Information Form, the Premenstrual Syndrome Scale (PMSS), and the WHOQOL-BREF-TR Quality of Life Scale. Data obtained in the study will be entered into a database using IBM SPSS 25.0 (Statistical Package for the Social Sciences), and all necessary statistical analyses will be conducted in the same program.

ELIGIBILITY:
Inclusion Criteria:

* Must be an undergraduate student studying midwifery at Istanbul University-Cerrahpaşa Faculty of Health Sciences.
* Must have a score of 110 or higher on the PMSS.
* Must have an internet connection.
* Must have the Zoom program installed and ready to use on their electronic device (phone or computer).

Exclusion Criteria:

* Must be under 18 years of age.
* Must have a change in menstrual cycle characteristics after being diagnosed with PMS.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
The Effect of Mandala Coloring on Premenstrual Syndrome Symptoms | eight weeks
  Premenstrual Syndrome Scale (PMSS): Developed by Gençdoğan in 2006, this five-point Likert-type scale measures the severity of premenstrual problems, consisting of 44 items and nine subscales. The lowest possible score is 44, and the highest is 220. A higher score indicates a greater severity of PMS problems.
The Effect of MMusic Listening on Premenstrual Syndrome Symptoms | eight weeks
  Premenstrual Syndrome Scale (PMSS): Developed by Gençdoğan in 2006, this five-point Likert-type scale measures the severity of premenstrual problems, consisting of 44 items and nine subscales. The lowest possible score is 44, and the highest is 220. A higher score indicates a greater severity of PMS problems.

SECONDARY OUTCOMES:
The Effect of Mandala Coloring Quality of Life | eight weeks
  WHOQOL-BREF-TR Quality of Life Scale: The Turkish version of the scale has been shown to be valid and reliable. The scale includes subdomains of physical health, psychological health, social relationships, and environment and culture-standardized environmental assessment. Each domain is scored between 4 and 20, with higher scores indicating higher quality of life in that area.
The Effect of Music Listening on Quality of Life | eight weeks
  WHOQOL-BREF-TR Quality of Life Scale: The Turkish version of the scale has been shown to be valid and reliable. The scale includes subdomains of physical health, psychological health, social relationships, and environment and culture-standardized environmental assessment. Each domain is scored between 4 and 20, with higher scores indicating higher quality of life in that area.

CONTACTS AND LOCATIONS:
Overall Officials: RUKIYE DUMAN, RESEARCH ASSISTANT, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University- Cerrahpasa, Istanbul, AVCILAR, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No